CLINICAL TRIAL: NCT01892761
Title: THE PROFILE OF MYCOPHENOLIC ACID IN CONSECUTIVE PHARMACOKINETICS AFTER RENAL TRANSPLANTATION:EFFECTS OF TIME AND CALCINEURIN-INHIBITORS
Brief Title: MPA Pharmacokinetics in Renal Transplantation
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAPPesq 1013/02
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Transplantation Recipients
Keywords: mycophenolate mofetil; mycophenolic acid; MPA; MMF; Pharmacokinetics; renal transplantation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TCL/MMF Group
  Interventions: Drug: Renal transplant recipients were allocated to TCL/MMF or to CyA/MMF groups
- CyA/MMF Group
  Interventions: Drug: Renal transplant recipients were allocated to TCL/MMF or to CyA/MMF groups

INTERVENTIONS:
Drug: Renal transplant recipients were allocated to TCL/MMF or to CyA/MMF groups

SUMMARY:
Adequate exposure to mycophenolic acid (MPA) is associated with better outcomes in kidney transplantation. This study evaluated repeated, MPA pharmacokinetics (MPA-PK) according to post-transplant time-points and concomitant CNIs. Fifty-two patients, 33 allocated to tacrolimus (TCL) and 19 to CyA (all with mycophenolate mofetil (MMF) and steroids), had the full MPA area under the time-concentration curve (AUC0-12hrs) repeatedly evaluated at days 7, 14, 30, 60 and 180 post-transplant. MMF daily dose was lower in TCL group as per protocol. Dose-adjusted MPA-AUC0-12hrs progressively increased throughout the study period in both groups but profiles were different according to the CNI regimen and time. The majority of patients were underexposed to MPA on day 7 for both groups what reinforces the need of a higher dose in the first week. Dose-adjusted MPA-AUC0-12hrs was higher in TCL group, after day 7, due to both a diminished MPA clearance (for both groups) and higher AUC4-12hrs in the TCL group. There was a progressive overexposure to MPA in order that at day 180, 21-30% of the patients were overexposed to MPA what indicates a time for MPA monitoring and dose correction for long-term follow-up. These PK data suggest that changes in MPA profile occur according to time and CNIs used and suggests that MPA monitoring may be mandatory at specific time-points.

ELIGIBILITY:
Male and female patients aged 18-65 years, recipients of a non-HLA identical kidney allograft who presented a PRA < 50% were eligible for the MoDIFY trial. Subjects were excluded if they received a non-renal organ, had current history of alcohol or illicit drug abuse, had liver enzymes more than two times the upper normal limit or received induction with anti-lymphocyte preparations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2002-09; Primary Completion 2003-03 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To establish the dynamics of MPA-PK (AUC0-12hrs) during the first six months | 6 months
  To establish the dynamics of MPA-PK during the first six months following transplantation according to time and the CNI regimen used in 52 patients who had their full MPA-PK monitored in 5 post-transplant time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Elias David-Neto, MD, PhD, Principal Investigator — Renal Transplantation Service - Hospital das Clínicas - University of São Paulo School of Medicine, Sao Paulo, Brazil
Locations (1):
- Renal Transplantation Service, São Paulo, São Paulo, Brazil